CLINICAL TRIAL: NCT06980935
Title: Individualized 130 Hz Subthalamic Temporal Interference Stimulation Versus Medication for Motor Symptoms in Parkinson Disease
Brief Title: STN-tTIS Modulates Parkinson Motor Symptoms With and Without Medications
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2025140A
Record Dates: First submitted 2025-05-11; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: subthalamic nucleus; transcranial temporal interference stimulation; MDS-UPDRS-Ⅲ
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Only use STN - tTIS therapy. (Experimental): Patients in this group received two 20-minute individualized 130 Hz STN-tTIS sessions targeting the more affected hemisphere's STN during medication "off" (≥12 hours withdrawal) and were evaluated for the MDS - UPDRS - III before and after treatment.
  Interventions: Device: NervioX-2400
- STN - tTIS therapy is used in combination with medication. (Experimental): Patients in this group received two 20-minute individualized 130 Hz STN-tTIS sessions targeting the more affected hemisphere's STN during medication "on" and were evaluated for the MDS - UPDRS - III before and after treatment.
  Interventions: Device: NervioX-2400

INTERVENTIONS:
Device: NervioX-2400 — To design the individualized tTIS, each participant completed a T1-weighted anatomical magnetic resonance imaging (MRI) scan. The individual's structural brain MRI data were used to determine the tTIS montage and stimulation settings via computational modeling.

SUMMARY:
The goal of this clinical trial is to evaluate the immediate effects of individualized 130 Hz STN-tTIS(Subthalamic Nucleus - transcranial Temporal Interference Stimulation)on motor symptoms in early-to-mid-stage PD patients during both medication "on" and "off" states. The main questions it aims to answer are:

1. Does the therapeutic effect of STN - tTIS relate to medication?
2. The degree of improvement in motor symptoms of Parkinson's disease patients after STN - tTIS therapy under different medication conditions.

Researchers compared the MDS - UPDRS - III improvement scores of tTIS therapy in the "on" and "off" medication phases to see if tTIS could work of independently medication.

1. Visit the clinic once every 1 weeks for therapy and test.
2. Record their symptoms and scores.

DETAILED DESCRIPTION:
This clinical trial aims to explore whether individualized 130 Hz subthalamic tTIS can improve motor symptoms of PD independently of medication. . Each participant underwent two separate 20-minute sessions of individualized 130 Hz STN-tTIS: one during medication "on" (defined as stable dopaminergic medication effect) and one during medication "off" (after ≥12 hours withdrawal of dopaminergic medications). The order of sessions was randomized with at least 7 days washout between sessions to avoid carryover effects. And MDS - UPDRS - III scales are assessed before and after each treatment.

ELIGIBILITY:
Inclusion Criteria:

* MDS diagnosis of primary Parkinson's disease
* Hoehn & Yahr stage < 3
* Antiparkinsonian drugs remained unchanged in the past four weeks and dosage remained unchanged during the study

Exclusion Criteria:

* Presence of neurological disorders that may affect the study (e.g., Traumatic brain injury)
* History of antipsychotics, antidepressants, or dopamine modulators other than PD drugs
* Metal devices in the head or heart (e.g., deep brain stimulators, pacemakers)
* Unstable vital signs

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-18 (Estimated)

PRIMARY OUTCOMES:
MDS-UPDRS-Ⅲ scores | pre-intervention, immediately after the intervention
  The score range for MDS-UPDRS-Ⅲ is from 0 to 132. Minimum Value: 0, indicating no motor impairment. Maximum Value: 132, indicating the most severe motor impairment.
  Higher scores on the MDS-UPDRS-Ⅲ indicate worse outcomes, as they reflect greater severity of motor symptoms.

SECONDARY OUTCOMES:
MDS-UPDRS-Ⅲ sub-scores | pre-intervention, immediately after the intervention
  The MDS-UPDRS-Ⅲ assesses motor symptoms in Parkinson's disease through sub-scores:
  Tremor Sub-score: Items 15-18; range 0-16. Higher scores indicate more severe tremors.
  Rigidity Sub-score: Item 3; range 0-12. Higher scores reflect greater rigidity. Bradykinesia Sub-score: Items 2, 4-9, and 14; range 0-40. Higher scores indicate more severe slowness of movement.
  Axial Sub-score: Items 1 and 9-13; range 0-24. Higher scores suggest more significant axial impairments.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China